CLINICAL TRIAL: NCT00243646
Title: Implant and External Radiation for Prostate Cancer With or Without Hormonal Therapy: A Prospective Randomized Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Schiffler Cancer Center (Other)
Collaborators: Kent E. Wallner, M.D. (Unknown); Sylvester, John, M.D. (Individual)
Responsible Party: Principal Investigator, Gregory Merrick, M.D., Medical Director, Schiffler Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-8-4
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Radiation therapy; Brachytherapy; Prostatic neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no hormones (Active Comparator): All patients will receive a 5-week course of external beam radiation therapy to the pelvis and a Pd-103 brachytherapy implant with no hormones
  Interventions: Radiation: External beam radiation
- 9 months of hormone therapy (Active Comparator): All patients will receive a 5-week course of external beam radiation therapy to the pelvis and a Pd-103 brachytherapy implant with a 9 month course of hormone therapy
  Interventions: Radiation: External beam radiation; Drug: Lupron; Drug: Casodex

INTERVENTIONS:
Radiation: External beam radiation — All patients will receive a 5-week course of external beam radiation therapy to the pelvis and a Pd-103 brachytherapy implant
Drug: Lupron — 9 months of an LHRH agonist and 4 months of an anti-androgen) is optimal for securing long-term biochemical control (a stable, non-rising PSA).
  Arms: 9 months of hormone therapy
Drug: Casodex — 9 months of an LHRH agonist and 4 months of an anti-androgen) is optimal for securing long-term biochemical control (a stable, non-rising PSA).
  Arms: 9 months of hormone therapy

SUMMARY:
Determine the role of androgen deprivation therapy in high risk patients receiving 45 Gy of pelvic radiotherapy plus a Pd-103 boost and the impact of the duration of ADT in hormonally-manipulated patients.

DETAILED DESCRIPTION:
In calender year 2005, 220, 000 men will be diagnosed with prostate cancer and approximately 30,000 will subsequently die of metastatic disease. Although the vast majority of men will be diagnosed with clinically localized and potentially curable disease, the selection of one local modality over another remains a focus of significant controversy within the uro-oncology community. However, patients with higher risk features are most often managed with radiotherapeutic approaches to include androgen deprivation therapy.

Prostate brachytherapy represents the ultimate-three dimensional conformal therapy and permits dose escalation far exceeding other modalities. Following permanent prostate brachytherapy with or without supplemental external beam radiation therapy, favorable long-term biochemical outcomes have been reported for patients with low, intermediate and high risk features with a morbidity profile that compares favorably with competing local modalities (1,2).

Several prospective randomized trials have demonstrated that androgen deprivation therapy in conjunction with conventional doses of external beam radiation therapy (65-70 Gy)results in improvement in disease-free and overall survival in patients with locally advanced prostate cancer (3,4).

ELIGIBILITY:
Inclusion Criteria:

* High risk patients - Two to three of the following: PSA 10-30 ng/mL, Gleason score greater than or equal to 6, clinical stage greater than or equal to T2c (2002 ACJJ).
* CT of the abdomen and pelvis and bone scan without evidence of metastases.
* An enzymatic prostatic acid phosphatase must be obtained prior to randomization.
* A serum testosterone must be obtained prior to initiation of androgen deprivation therapy.
* No prior pelvic external beam radiation therapy for prostate cancer or other malignancies.
* No prior androgen deprivation therapy.
* Minimum 5 year life expectancy.
* No other invasive cancer diagnosis other than non-melanoma skin cancer within the last 5 years.

Exclusion Criteria:

* Exclusion criteria will be limited to patients who do not meet the above eligibility criteria.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
PSA 3 and 6 months following implantation then every 6 months. | 3 and 6 months following implantation then every 6 months
  PSA 3 and 6 months following implantation then every 6 months.
Serum testosterone levels at 3 and 6 months in hormonally manipulated patients. | 3 and 6 months
  Serum testosterone levels at 3 and 6 months in hormonally manipulated patients
Androgen deprivation therapy will not be reinitiated unless the post-treatment PSA exceeds 10 ng/mL or distant metastases are detected. | as needed
  Androgen deprivation therapy will not be reinitiated unless the post-treatment PSA exceeds 10 ng/mL or distant metastases are detected.

SECONDARY OUTCOMES:
EPIC on 6 and 12 months and then annually. | 6 and 12 months and then annually.
  EPIC on 6 and 12 months and then annually.
Hormonally manipulated patients will obtain a DEXA scan. | as needed
  Hormonally manipulated patients will obtain a DEXA scan.
For documented osteoporosis, Zometa (4 mg IV over 15 minutes) every 3 months is recommended. | every 3 months is recommended.
  For documented osteoporosis, Zometa (4 mg IV over 15 minutes) every 3 months is recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S Merrick, MD, Principal Investigator — Schiffler Cancer Center, Wheeling, WV; Kent E. Wallner, MD, Study Chair — Group Health Cooperative, Veterans Administration Hospital, and University of Washington; John Sylvester, MD, Study Chair — Seattle Prostate Institute Seattle, WA 98104
Locations (3):
- United States (3):
  - Seattle Prostate Institute, Seattle, Washington
  - Groupe Health Cooperative, Veterans Adminstration Hospital and University of Washington, Seattle, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia

REFERENCES:
- [Background] Merrick GS, Wallner KE, Butler WM. Permanent interstitial brachytherapy for the management of carcinoma of the prostate gland. J Urol. 2003 May;169(5):1643-52. doi: 10.1097/01.ju.0000035544.25483.61. PMID 12686802
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Pilepich MV, Caplan R, Byhardt RW, Lawton CA, Gallagher MJ, Mesic JB, Hanks GE, Coughlin CT, Porter A, Shipley WU, Grignon D. Phase III trial of androgen suppression using goserelin in unfavorable-prognosis carcinoma of the prostate treated with definitive radiotherapy: report of Radiation Therapy Oncology Group Protocol 85-31. J Clin Oncol. 1997 Mar;15(3):1013-21. doi: 10.1200/JCO.1997.15.3.1013. PMID 9060541
- [Background] Roach M 3rd, DeSilvio M, Lawton C, Uhl V, Machtay M, Seider MJ, Rotman M, Jones C, Asbell SO, Valicenti RK, Han S, Thomas CR Jr, Shipley WS; Radiation Therapy Oncology Group 9413. Phase III trial comparing whole-pelvic versus prostate-only radiotherapy and neoadjuvant versus adjuvant combined androgen suppression: Radiation Therapy Oncology Group 9413. J Clin Oncol. 2003 May 15;21(10):1904-11. doi: 10.1200/JCO.2003.05.004. PMID 12743142
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Crook J, Ludgate C, Malone S, Lim J, Perry G, Eapen L, Bowen J, Robertson S, Lockwood G. Report of a multicenter Canadian phase III randomized trial of 3 months vs. 8 months neoadjuvant androgen deprivation before standard-dose radiotherapy for clinically localized prostate cancer. Int J Radiat Oncol Biol Phys. 2004 Sep 1;60(1):15-23. doi: 10.1016/j.ijrobp.2004.02.022. PMID 15337535
- [Background] Merrick GS, Butler WM, Galbreath RW, Lief JH, Adamovich E. Does hormonal manipulation in conjunction with permanent interstitial brachytherapy, with or without supplemental external beam irradiation, improve the biochemical outcome for men with intermediate or high-risk prostate cancer? BJU Int. 2003 Jan;91(1):23-9. doi: 10.1046/j.1464-410x.2003.04024.x. PMID 12614244
- [Background] Merrick GS, Butler WM, Wallner KE, Galbreath RW, Lief JH, Allen Z, Adamovich E. Impact of supplemental external beam radiotherapy and/or androgen deprivation therapy on biochemical outcome after permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):32-43. doi: 10.1016/j.ijrobp.2004.05.003. PMID 15629591
- [Background] Lee LN, Stock RG, Stone NN. Role of hormonal therapy in the management of intermediate- to high-risk prostate cancer treated with permanent radioactive seed implantation. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):444-52. doi: 10.1016/s0360-3016(01)02598-6. PMID 11872291
- [Background] Stock RG, Cahlon O, Cesaretti JA, Kollmeier MA, Stone NN. Combined modality treatment in the management of high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2004 Aug 1;59(5):1352-9. doi: 10.1016/j.ijrobp.2004.01.023. PMID 15275720
- [Background] Sylvester J, Blasko JC, Grimm PD, Meier R, Goy B, Colburn G, Cavanagh W. Neoadjuvant Androgen Ablation Combined with External-Beam Radiation Therapy and Permanent Interstitial Brachytherapy Boost in Localized Prostate Cancer. Mol Urol. 1999;3(3):231-236. PMID 10851328
- [Background] Merrick GS, Butler WM. Modified uniform seed loading for prostate brachytherapy: rationale, design, and evaluation. Tech Urol. 2000 Jun;6(2):78-84. PMID 10798804
- [Background] Consensus statement: guidelines for PSA following radiation therapy. American Society for Therapeutic Radiology and Oncology Consensus Panel. Int J Radiat Oncol Biol Phys. 1997 Mar 15;37(5):1035-41. No abstract available. PMID 9169810
- [Background] Wallner K, Merrick G, True L, Sutlief S, Cavanagh W, Butler W. 125I versus 103Pd for low-risk prostate cancer: preliminary PSA outcomes from a prospective randomized multicenter trial. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1297-303. doi: 10.1016/s0360-3016(03)01448-2. PMID 14630265
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727